CLINICAL TRIAL: NCT00267176
Title: A 4-week, Multicentre, Randomized, Double-blind, Double-dummy, Parallel Group Ambulatory Blood Pressure Monitoring Study to Investigate Whether Treatment With Lumiracoxib 100 mg Once Daily Results in an Improved 24-hour Blood Pressure Profile Compared to Ibuprofen 600 mg Three Times a Day in Osteoarthritis Patients With Controlled Hypertension
Brief Title: Safety and Efficacy of Lumiracoxib in Patients With Osteoarthritis and With Controlled Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCOX189A2428
Record Dates: First submitted 2005-12-16; First posted 2005-12-20 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Osteoarthritis; Controlled Hypertension
Keywords: Osteoarthritis,; hypertension,; lumiracoxib,; ibuprofen,; 24-hour blood pressure profile
MeSH Terms: conditions — Osteoarthritis; Hypertension | interventions — lumiracoxib

INTERVENTIONS:
Drug: lumiracoxib

SUMMARY:
This study will investigate the effect on ambulatory blood pressure of lumiracoxib 100 mg once daily versus ibuprofen 600 mg three times a day in osteoarthritis patients with controlled hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the hand, hip, knee or spine
* High blood pressure (<140/ 90 mmHg) which is controlled by antihypertensive medication(s).

Exclusion criteria

• Evidence or history of any cardiac and cerebral thrombotic/ ischemic diseases and/ or events

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 1020
Dates: Start 2005-11; Primary Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Assessment of the 24-hour systolic BP profile of lumiracoxib 100 mg o.d. in comparison to ibuprofen 600 mg t.i.d. after 4 weeks of treatment.

SECONDARY OUTCOMES:
Assessment of the effect of lumiracoxib 100 mg o.d. on diastolic BP derived from ABPM after 4 weeks of treatment in comparison to ibuprofen 600 mg t.i.d.
Assessment of the effect of lumiracoxib 100 mg o.d. on daytime and nighttime BP (systolic and diastolic) derived from ABPM after 4 weeks of treatment in comparison to ibuprofen 600 mg t.i.d.
Assessment of the effect of lumiracoxib 100 mg o.d. on the incidence of significant increases in ABP in comparison to ibuprofen 600 mg t.i.d.
Exploratory analysis of the effect of lumiracoxib 100 mg o.d. on the incidence of uncontrolled hypertension in comparison to ibuprofen 600 mg t.i.d.
Exploratory analysis of the effect of lumiracoxib 100 mg o.d. on the ABPM profile between 0 and 4 hours after morning dose in comparison to ibuprofen 600 mg t.i.d.

CONTACTS AND LOCATIONS:
Overall Officials: Bradkey Sakran, MD, Principal Investigator — Southern Illinois Clinical Research
Locations (2):
- Southern Illinois Clinical Research, O'Fallon, Illinois, United States
- Novartis, Nuremberg, Germany

REFERENCES:
- [Result] MacDonald TM, Reginster JY, Littlejohn TW, Richard D, Lheritier K, Krammer G, Rebuli R. Effect on blood pressure of lumiracoxib versus ibuprofen in patients with osteoarthritis and controlled hypertension: a randomized trial. J Hypertens. 2008 Aug;26(8):1695-702. doi: 10.1097/HJH.0b013e328302c9fe. PMID 18622250